CLINICAL TRIAL: NCT03612024
Title: Next of Kin Survey Following Organ Donation Request - a Single Center Experience
Brief Title: Bernese Next of Kin Survey Following Organ Donation Request
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Principal Investigator, Andreas Bloch, Andreas Bloch, MD, Concultant Intensive Care Medicine, Insel Gruppe AG, University Hospital Bern
Other Study IDs: BNoKSurvey FODR
Record Dates: First submitted 2018-07-24; First posted 2018-08-02 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Organ Donation; Next of Kin; Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- request for organ donation approved
  Interventions: Behavioral: questionnaire
- request for organ donation rejected
  Interventions: Behavioral: questionnaire

INTERVENTIONS:
Behavioral: questionnaire — a standardized questionnaire was sent to all participants

SUMMARY:
6 to 18 months after organ donation request a next of kin survey using a standardized questionnaire was conducted.

ELIGIBILITY:
Inclusion Criteria:

Next of kin involved in request for organ donation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Next of kin involved in request for organ donation. Single center study. The request for organ donation must have passed 6 to 18 months ago
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-24 (Actual)

PRIMARY OUTCOMES:
factors influencing approval/rejection of an organ donation | 6 to 18 months pre questionnaire
factors with influence on mourning porcess | 6 to 18 months past request

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Bloch, MD, Principal Investigator — department of critical care medicine, inselspital, university hospital, bern, university of bern
Locations (1):
- Department for Intensive Care Medicine, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nebiker M, Bloch A, Fedakar P, Christen L, Hurni A, Carre D, Cluzet S, Eckert P, Schefold JC. Organ donation in the ICU - a survey on next of kin response in two Swiss academic centres. Swiss Med Wkly. 2021 Jun 23;151:w20515. doi: 10.4414/smw.2021.20515. eCollection 2021 Jun 21. PMID 34161597